CLINICAL TRIAL: NCT06373939
Title: Pivotal Study of the Performance and Safety of the Pneumoscope Device in Adults and Children
Brief Title: Performance and Safety of the Pneumoscope Device in Adults and Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pneumoscope study
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Diseases; Pneumonia; Asthma; Cyanotic Heart Disease
Keywords: Stethoscopes; Oxygen Saturation; Thermometers; Digital Health; Auscultation
MeSH Terms: conditions — Respiratory Tract Diseases; Pneumonia; Asthma | interventions — Thermometers

STUDY DESIGN:
Intervention Model Description: This single center, open, non-controlled investigation will be conducted at one site; the University Hospitals of Geneva, Switzerland. This will be a non-inferiority study between Pneumoscope and CE marked comparable medical devices in children and adults.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children (>1 year old) and adult patients (Experimental): Patients with various respiratory conditions, such as asthma or pneumonia, along with healthy individuals, will be targeted to assess the Pneumoscope's performance under clinical conditions. Additionally, patients with lower blood oxygen saturation levels, such as those with cyanotic heart defects like tetralogy of Fallot, will also be included
  Interventions: Device: Digital lung auscultation; Device: Pulse oximetry measurement; Device: Non invasive body temperature measurement

INTERVENTIONS:
Device: Digital lung auscultation — Two 30-second recordings will be made using CE-marked Littmann® CORE digital stethoscopes and the Pneumoscope at two bilateral lung positions on the posterior chest wall, focusing on the lower lobes. Spectral comparison and audio quality indices will be assessed between the Pneumoscope and the Littmann® CORE digital stethoscope.
  Comparator: The Gold Standard Littmann® CORE picks up sounds, such as heart and lung sounds, from a patient's body. After amplification and filtering, the sounds are sent to the user through a binaural headset. The stethoscope chest piece is designed for use with adult, pediatric, and infant patients.
Device: Pulse oximetry measurement — Pulse oximetry and heart rate will be measured using the CE-marked Masimo Rad-G® and iHealth® Air oximeters, as well as the Pneumoscope's built-in oximeter. Agreement between the Pneumoscope's oximeter and the reference oximeters will be evaluated. Measurement will take 30 second on the right index finger.
  Comparators:
  1. The Gold Standard Masimo Rad-G® sensor is indicated for the continuous noninvasive peripheral monitoring of arterial oxygen saturation (SpO2) and pulse rate. Its use consists in positioning the emitting window of the sensor attachment envelope on the top of the finger nail bed, while the detector is placed opposite the emitter on the other side of the same finger.
  2. The Gold Standard iHealth® Air works by projecting two beams of light through a clip with a transmitter and a detector that is placed around a finger, nail side down and screen side up.
  Other Names: Oximeters
Device: Non invasive body temperature measurement — Comparison of body temperature measurements between the Pneumoscope's built-in thermometer and Gold Standard thermometers (Terumo® C205 and VisioFocus Pro 06480).
  Comparators:
  1. The Gold Standard Terumo® C205 is an axillary thermometer. Its use consists in placing the probe in the armpit, then lowering the arm and holding the device firmly until the temperature is stabilised and the temperature is read and displayed on the thermometer screen.
  2. The Gold Standard VisioFocus Pro 06480 is an infrared thermometer that detects the infrared radiation naturally emitted by the body and in particular from the human forehead. Its use consists in holding the thermometer close to the forehead but without direct contact with the skin. The temperature reading is then projected on the patient's forehead using a symbol system.
  Other Names: Thermometers

SUMMARY:
Respiratory diseases are associated with high morbidity and mortality worldwide. Proper diagnosis and risk assessment of these conditions are essential for optimal management. Clinicians use three particularly useful tools to identify these conditions when assessing the patient's status: the stethoscope, the pulse oximeter, and the thermometer. The Pneumoscope is an all-in-one device including a digital stethoscope, a pulse oximeter, and a thermometer. This study aims to assess the performance and safety of the Pneumoscope in recording respiratory sounds, body temperature, non-invasive blood oxygen saturation levels and heart rate in children and adults.

DETAILED DESCRIPTION:
Respiratory diseases affect over 500 million people globally, ranking third in causes of death. Chronic obstructive pulmonary diseases impact 251 million individuals due to air pollution and tobacco smoke. Asthma is the most prevalent chronic disease in children, while pneumonia is the leading cause of death in children under 5. Respiratory infections are prominent in pediatric outpatient clinics, especially in low- and middle-income countries. Accurate diagnosis and risk assessment are crucial for effective management. Clinicians utilize three key tools: the stethoscope for auscultation, detecting abnormal breathing sounds; the pulse oximeter, indicating oxygen deficiency in inflamed lungs; and the thermometer, primarily for fever-related infections like pneumonia. Auscultation, while quick and non-invasive, suffers from user-dependent subjective interpretation, as highlighted by studies reporting low correct response rates, especially among non-pulmonologists. Pulmonary auscultation's sensitivity and specificity are notably low, particularly in unilateral or focal changes. Pulse oximetry, utilizing harmless light wavelengths, measures oxygenated hemoglobin concentration, with a saturation below 92% indicating hypoxia, albeit with reduced accuracy below 90%. Thermometers measure body temperature, with rectal measurement considered the gold standard in children, although non-contact methods remain contentious

The use of the Pneumoscope, a digital medical device, could address the above challenge. The Pneumoscope is designed to enhance respiratory disease diagnosis and provide heart rate, respiratory rate, pulse oximetry, and body temperature data. This project aims to evaluate its performance against gold standards in lung sound processing, pulse oximetry, and body temperature measurement. Furthermore, the Pneumoscope is envisioned to integrate artificial intelligence (AI) for future applications. Data on breath sounds, oximetry, heart rate, and temperature from patients with respiratory diseases will inform AI algorithms for disease recognition and risk assessment. Ultimately, this technology could enable remote diagnosis and follow-up, particularly beneficial for patients in low- and middle-income countries or with limited mobility. However, the current study focuses solely on assessing the Pneumoscope's performance as a standard digital stethoscope with integrated temperature and oximetry sensors, aiming to establish agreement with established clinical tools for digital lung auscultation, pulse oximetry, heart rate, and body temperature measurement.

This is a single center, open, non-controlled investigation that will be conducted at the University Hospitals of Geneva, Switzerland. This will be a non-inferiority study between Pneumoscope and CE marked comparable medical devices in children and adults.

ELIGIBILITY:
Patients will be recruited from the pediatric and adult clinical departments of the Geneva University Hospitals.

Inclusion Criteria:

* Age > 1 year old.
* Healthy patients on the day of auscultation OR
* Patients with lower respiratory tract diseases (e.g., bronchitis, pneumonia, etc.). OR
* Patients with low (i.e., <92%) pulse oximetry values (e.g., cyanotic heart defect such as tetralogy of Fallot, transposition of great vessels, etc.). AND / OR
* Patients with fever >38.0°C.
* And for all: Information and written consent of the patient or a legal representative.

Exclusion Criteria:

* Refusal of consent.
* Clinical signs of severity: acute hypoxia, hypercapnia, acute respiratory failure, acute circulatory failure.
* Immune disorder, primary ciliary dyskinesia, antecedent of neonatal bronchopulmonary dysplasia.
* Contraindications and limitations of the MD as described in the instructions for use.
* Contraindications to the class of medical devices being studied, e.g. known hypersensitivity or allergy to the device material.
* Clinically significant concomitant disease states.
* Inability to follow the study procedures, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another study with an investigational drug or other medical device within 30 days prior to and during the present study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Pneumoscope's built-in sensors | During procedure, i.e. 20 minutes per patient for both out- and inpatients.
  To be used in patients and certified by competent authorities the performance of Pneumoscope has to be at least equal as comparable devices on the market. Performances of digital audio quality, as well as pulse oximetry, heart rate and temperature measurements by the Pneumoscope will be compared to CE certified similar medical devices used as gold-standards tools. Hence, the primary objective is to evaluate whether the three built-in sensors into the Pneumoscope are equivalent to CE marked Gold Standards:
  1. Spectral comparison and other audio quality indices of recordings with the Pneumoscope and a commercially available digital stethoscope (Littmann® CORE digital stethoscope).
  2. Agreement between the Pneumoscope thermometer and reference thermometers (Terumo® C205 and VisioFocus Pro® 06480).
  3. Agreement between the Pneumoscope pulse oximeter (for blood oxygen saturation and heart rate) and reference oximeters (Masimo Rad-G® and iHealth® Air).

SECONDARY OUTCOMES:
Collect audio records of lung sounds for AI models training and sensor calibration | During procedure, i.e. 20 minutes per patient for both out- and inpatients.
  The collected anonymised audio records of lung sounds will be used in the future to develop and validate AI algorithms for various bronchopulmonary diseases in children (pneumonia, asthma, bronchiolitis), as well as SARS-CoV-2 infections in adults.
Pulse oximetry | During procedure, i.e. 20 minutes per patient for both out- and inpatients.
  The collected pulse oximetry measures will be used to calibrate the oximeter sensor.
Body temperature | During procedure, i.e. 20 minutes per patient for both out- and inpatients.
  The collected, non-invasive, body temperature measures will be used to calibrate the thermometer sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Gervaix, Prof, Study Director — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
* Data types: Deidentified participant data. The final database will be shared on a non-commercial repository following the FAIR data principles.
  * How to access data: contact the principal investigator Dr Johan N. Siebert at: Johan.Siebert@hcuge.ch
  * When available: beginning 6 months and ending 10 years following article(s) publication.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 10 years following article(s) publication
Access Criteria: * Who can access the data: Data will be made available to qualified external researchers whose proposed use of the data has been approved by their Institutional Review Board.
  * Types of analyses: Data will be made available for a specified research purpose.
  * Mechanisms of data availability: Data will be made available upon approval of a proposal and with a signed data access agreement.
  * Any additional restrictions: The request proposal must include a statistician.